CLINICAL TRIAL: NCT02928185
Title: Adaptation of Coping Together, Self-directed Coping Skills Training Manuals for Patients and Caregivers in the Context of Hematopoietic Stem Cell Transplantation
Brief Title: Adaptation of Skills Training Manuals for Patients Receiving Hematopoietic Stem Cell Transplantation and Their Caregivers
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: City University of New York (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1334
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Post Hematopoietic Stem Cell Transplantation
Keywords: training manuals; patients and caregivers; 16-1334

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- HSCT patients: Individual/dyadic semi-structured interviews between Day +100 to +130
  Interventions: Behavioral: semi-structured interviews
- HSCT care givers: Individual/dyadic semi-structured interviews between Day +100 to +130
  Interventions: Behavioral: semi-structured interviews
- HSCT dyads: Individual/dyadic semi-structured interviews between Day +100 to +130
  Interventions: Behavioral: semi-structured interviews
- HSCT Clinicians: Can include: MD, RN, SW, PharmD and Nutritionist. Individual semi-structured interviews after 14 days to review the Coping Together manuals
  Interventions: Behavioral: semi-structured interviews

INTERVENTIONS:
Behavioral: semi-structured interviews

SUMMARY:
The purpose of this study is to see what the patients perceptions are of the Coping Together manuals during the first 100 days after their Hematopoietic Stem Cell Transplantation (HSCT), and if they would make any changes to Coping Together manuals for future patients, caregivers and couples that use these manuals after their HSCT. The investigators would also like to see what is the caregiver's perception of this intervention, and to see if they have any suggestions for changes. If the caregiver is interested in providing feedback, they will sign a separate consent form.

DETAILED DESCRIPTION:
A two-part, qualitative descriptive design will be employed to systematically adapt the Coping Together manuals based on recommendations of HSCT patients, CGs, dyads and clinicians (for Phase 1 only). For this study, CG is defined as spouse, partner, family member, friend, colleague, or neighbor who can, but do not necessarily live together, and provide uncompensated care. A dyad is defined as a combination of a patient and their designated CG. Dyads can review the Coping Together manuals individually or jointly, but will be interviewed together.

Part 1 will capture diverse perspectives of HSCT patients, CGs, dyads and clinicians using individual (patients, CGs, clinicians) and dyadic (dyads) interviews for the preliminary adaptation of the Coping Together manuals.

Part 2 will explore the experiences of HSCT patients, CGs and dyads with HSCT CT, which will be the HSCT-modified version of the Coping Together manuals, using individual (patients, CGs) and dyadic (dyads) interviews to refine the HSCT CT manuals.

ELIGIBILITY:
Inclusion Criteria:

Part 1

HSCT Patients

* Admission to the MSKCC Adult BMT service for an outpatient HSCT for a hematologic malignancy
* HSCT procedure scheduled within two months of consent
* ≥18 years old
* Ability to read, speak and understand English
* Able to give written informed consent
* Physically and cognitively able to participate in the study as determined by the investigators HSCT CGs
* ≥18 years old
* Ability to read, speak and understand English
* Able to give written informed consent
* Physically and cognitively able to participate in the study as determined by the investigators

HSCT Dyads

* In addition to meeting the inclusion criteria for HSCT Patients and HSCT CGs above, both parties must provide mutual agreement to participate as a dyad.

HSCT Clinicians

* Member of MSKCC BMT patient care team for at least one year

Part 2

HSCT Patients

* Same as Part 1 HSCT Patients HSCT CGs
* Same as Part 1 HSCT CGs HSCT Dyads
* Same as Part 1 HSCT Dyads

Exclusion Criteria:

Part 1 HSCT Patients

* Physically and cognitively unable to participate in the study as determined by the investigators HSCT CGs
* Inability to complete role responsibilities 24 hours per day for at least 50% of time (50 days)
* Physically and cognitively unable to participate in the study as determined by the investigators HSCT Dyads
* Participants must not meet the exclusion criteria for HSCT Patients and HSCT CGs above.
* Patients or CGs who are participating in this study as individuals HSCT Clinicians
* There are no exclusion criteria

Part 2 HSCT Patients

* Same as Part 1 HSCT Patients HSCT CGs
* Same as Part 1 HSCT CGs HSCT Dyads
* Same as Part 1 Dyads

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hematopoietic Stem Cell Transplantation and Their Caregivers at MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
finalize the preliminary adaptation of the manuals | 1 year
  Socio-demographic characteristics will be summarized with descriptive statistics (frequencies, percentages, means, standard deviations) using IBM SPSS® Statistics, Version 22.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Son, BS, MS, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Son T, Lambert S, Jakubowski A, DiCicco-Bloom B, Loiselle CG. Adaptation of Coping Together - a self-directed coping skills intervention for patients and caregivers in an outpatient hematopoietic stem cell transplantation setting: a study protocol. BMC Health Serv Res. 2018 Aug 29;18(1):669. doi: 10.1186/s12913-018-3483-1. PMID 30157867
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/